CLINICAL TRIAL: NCT01566799
Title: Clinical Phase II, Randomized, Double Blind Trial, to Evaluate the Efficacy of Metformin and Chemotherapy Versus Placebo Nad Chemotherapy in Neoadjuvant Setting for Locally Advanced Breast Cancer
Brief Title: Metformin Plus Neoadjuvant Chemotherapy in Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Collaborators: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Claudia Arce Salinas, Medico Especialista, Instituto Nacional de Cancerologia de Mexico
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MET-INCAN-1
Record Dates: First submitted 2012-03-22; First posted 2012-03-29 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Locally Advanced Malignant Neoplasm
Keywords: Locally advanced breast cancer; Neoadjuvant chemotherapy; Metformin; Pathologic Complete Response
MeSH Terms: conditions — Pathologic Complete Response | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): Patients will be receive 12 weeks of paclitaxel followed by 4 cycles of FAC combined with 500 mg/day of metformin p.o.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — metformin 500 mg/day po for 24 weeks.
  Other Names: Dabex

SUMMARY:
Background Obesity and overweight are well known risk factors for breast cancer and also are associated with higher recurrence and mortality rates.

Main goal of this study is to evaluate the efficacy of metformin plus chemotherapy in terms of pathologic complete response in comparison with placebo plus the same chemotherapy regimen Design: Randomized, double blind, clinical trial. This study will be performed at National Cancer Institute of Mexico City, at breast cancer unit.

Patients with ER+ or PR+, HER2 negative, breast cancer are candidates to participate.

After completion of chemotherapy all patients will have a breast surgery to assess pathologic response.

Complete pathologic response is defined as the abscence of malignant cells in breast tissue and lymph nodes. The presence of DCIS is considered as pCR

DETAILED DESCRIPTION:
Definitions Luminal A: tumors ER + PR + HER2 Negative and Ki67 <14% Luminal B: tumors ER +/-, PR +/-, HER2 negative and Ki67 >15% Complete pathologic response is defined as the abscence of malignant cells in breast tissue and lymph nodes. The presence of DCIS is considered as pCR

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 years old and younger than 70 years old

  * Invasive breast cancer confirmed by core biopsy, any histology
  * Tumor ≥2 cm and/or lymph node positive (proven by FNA)(T2-4b, N0-3, M0)
  * Must have ER/PR positive and HER2 negative
  * Must have full staging and extent disease and clinically and radiographically tumor measure
  * Without previous treatment for breast cancer (including surgery, hormonotherapy or chemotherapy)
* Normal liver, kidney and blood tests
* Performance Status ECOG 0-2 o Karnofsky ≥70%
* Fasten glucose levels <125 mg/dl
* Signed consent

Exclusion Criteria:

* Previous use of metformin for any indication
* Presence of Diabetes Mellitus

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response | pCR will be assesed after 24 weeks of treatment
  to assess the efficacy in terms of pahtologic complete response in patients with locally advanced breast cancer, treated with neoadjuvant chemotherapy based on Paclitaxel followed by FAC, combined with metformin or placebo

SECONDARY OUTCOMES:
Safety analysis | after 24 treatment weeks'
  For safety analysis we are going to use NCTC criteria version 3.0
Assess clinical response at the end of paclitaxel and at the end of neoadjuvant chemotherapy | after 24 treatment weeks'
  tumor measurements by caliper every cycle and by ultrasound at the end of chemotherapy
To correlate serum levels of insulin, protein C and HbA1 (after treatment) with clinical and pathologic response | safter 24 treatment weeks'
  correlation between serum levels of insuline levels, HbA1 and PCR and PCR

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Arce, MD, MSc, Principal Investigator — Instituto Nacional Canerologia
Locations (1):
- Instituto Nacional Cancerologi, Mexico City, Mexico City, Mexico